CLINICAL TRIAL: NCT02693314
Title: Evaluation of Jarro-Dophilus EPS® Probiotic Formulations on Probiotic Survival, Fecal Microbiota, Gastrointestinal Function and General Wellness in Healthy Adults: a Randomized, Double-blind, Dose-response Study
Brief Title: Evaluation of Jarro-Dophilus EPS® Probiotic Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201401031
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Jarro-Dophilus; probiotic; microbiota; gastrointestinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jarro-Dophilus EPS® Group (Experimental): Jarro-Dophilus EPS® (5 billion CFU/capsule) probiotic formulation capsule for 28 days
  Interventions: Dietary Supplement: Jarro-Dophilus EPS® (5 billion CFU/capsule)
- Jarro-Dophilus EPS® High Potency Group (Experimental): Jarro-Dophilus EPS® High Potency (25 billion CFU/capsule) probiotic formulation capsule for 28 days
  Interventions: Dietary Supplement: Jarro-Dophilus EPS® High Potency (25 billion CFU/capsule)
- Placebo Group (Placebo Comparator): Placebo capsule for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Jarro-Dophilus EPS® (5 billion CFU/capsule) — One capsule containing 5 billion CFU of the probiotic mix (Lactobacillus helveticus, Lactobacillus rhamnosus, Lactobacillus casei, Pediococcus acidilactici, Bifidobacteria breve, Bifidobacteria longum, Lactobacillus plantarum and Lactobacillus lactis ssp. lactis) will be taken once a day for a period of 28 days.
  Arms: Jarro-Dophilus EPS® Group
Dietary Supplement: Jarro-Dophilus EPS® High Potency (25 billion CFU/capsule) — One capsule containing 25 billion CFU of the probiotic mix (Lactobacillus helveticus, Lactobacillus rhamnosus, Lactobacillus casei, Pediococcus acidilactici, Bifidobacteria breve, Bifidobacteria longum, Lactobacillus plantarum and Lactobacillus lactis ssp. lactis) will be taken once a day for a period of 28 days.
  Arms: Jarro-Dophilus EPS® High Potency Group
Dietary Supplement: Placebo — One capsule (containing potato starch, magnesium stearate and ascorbic acid) will be taken once a day for a period of 28 days.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine the effects of the two doses of Jarro-Dophilus EPS® probiotic supplements on fecal lactobacillus and bifidobacteria numbers, transit survival of administered probiotic strains, fecal microbiota, gastrointestinal function and general wellbeing in healthy human adults.

DETAILED DESCRIPTION:
Participants will be screened using the International Physical Activity Questionnaire (questions regarding physical activity, including intensity, duration and frequency) and inclusion/exclusion criteria. Participants will be scheduled to begin a 7-day baseline period, during which participants will complete daily questionnaires of bowel movement frequency, gastrointestinal symptoms and wellness. On or about day 8, height and weight will be determined. Participants will then be randomized to one of the following groups:

Group 1: Jarro-Dophilus EPS® (5 billion CFU/capsule), Group 2: Jarro-Dophilus EPS® Higher Potency (25 billion CFU/capsule), Group 3: Placebo capsule

Study participants will continue to complete the daily online questionnaire throughout the 28 days of treatment and for 7 days post treatment. Participants will also be asked to complete a weekly questionnaire on gastrointestinal symptoms (Gastrointestinal Symptom Rating Scale) throughout the entire study. In addition, participants in each group will be asked to collect one stool sample at baseline, one stool sample during week 4 of treatment and an additional sample during the washout period. Stool samples will be analyzed and quantified for the probiotic bacteria and changes in the microbiota.

Participants will be asked to return any unconsumed supplements at the end of the treatment period. Additionally, the participants will be weighed after the treatment period and the washout period.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study you must

* be between18-50 years of age
* be willing to have your height and weight measured and provide demographic information
* be willing to consume a probiotic or placebo capsule daily for 4 weeks
* be willing to provide 3 stool samples during the study
* be willing to complete a daily questionnaires regarding general and gastrointestinal wellness and the Gastrointestinal Symptom Rating Scale weekly throughout the entire 6-wk study
* have daily access to a computer with Internet access for the entire 6-wk study
* be willing and able to provide a valid social security for study payment purposes
* be willing and able to provide a valid social security for study payment purposes
* be willing to complete the International Physical Activity Questionnaire (asks you to report physical activity including intensity, duration and frequency)

Exclusion Criteria:

To participate in the study you must NOT

* be currently taking medications for constipation or diarrhea
* have previously or are you currently being treated for any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's, Celiac, ulcerative colitis, etc.), other chronic diseases (diabetes, kidney disease, etc.) or immune-compromising diseases or conditions (HIV, AIDS, autoimmune, hepatitis, cancer, transplant patient etc.)
* have any known allergy to milk, milk protein, soy, gluten or have gluten sensitivity
* have taken antibiotics within the past 4 weeks prior to randomization
* be currently taking a probiotic supplement and are unwilling to discontinue it a minimum of 2 weeks prior to the study start
* be a current smoker.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Microbiota Studies (Composition) | Changes from Baseline, Week 4 of Treatment and Week 5
  Changes in fecal lactobacilli and bifidobacteria between treatment groups.

SECONDARY OUTCOMES:
Digestive Health (Bowel Movement Frequency) | Changes from Baseline at Week 1,2,3,4 and Week 5
  Bowel movement frequency will be self-reported using a daily questionnaire.
Digestive Health (Gastrointestinal Symptom Rating Scale) | Changes from Baseline at Week 1,2,3,4 and Week 5
  Measured by gastrointestinal symptoms (bloating, reflux, constipation, diarrhea) using the weekly Gastrointestinal Symptom Rating Scale (GSRS).
Digestive Health (Gastrointestinal Function and General Wellness) | Changes from Baseline at Week 1,2,3,4 and Week 5
  Measured by gastrointestinal symptoms (gas, bloating, diarrhea, etc) assessed using a daily questionnaire. The daily questionnaire will also include questions regarding wellness and the Bristol Stool Scale (stool form and transit).
Microbiota Studies (Recovery) | Changes from Baseline, Week 4 of Treatment and Week 5
  Change in the concentration and survival of the probiotic strains through intestinal passage using qPCR.
Microbiota Studies (Overall Composition) | Changes from Baseline, Week 4 of Treatment and Week 5
  Effects of the probiotic interventions on overall microbiota composition will be measured (e.g. 16S rRNA (ribosomal ribonucleic acid) sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided